CLINICAL TRIAL: NCT01323101
Title: Effect of Doxycycline on Sputum Biomarkers of Inflammation and Lung Epithelial Repair in Patients With Cystic Fibrosis.
Brief Title: Doxycycline Effects on Inflammation in Cystic Fibrosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Paul Beringer, Associate Professor, University of Southern California
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS-08-00017
Record Dates: First submitted 2011-02-15; First posted 2011-03-25 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): No doxycycline
  Interventions: Other: No doxycycline
- Doxycycline (Experimental)
  Interventions: Drug: Doxycycline

INTERVENTIONS:
Drug: Doxycycline — Doxycycline 40mg, 100mg, 200mg tablet once daily, or no drug for 28 days.
  Other Names: Doryx; Vibramycin
  Arms: Doxycycline
Other: No doxycycline
  Arms: Control

SUMMARY:
Doxycycline is known to exhibit immune modulatory activities beyond its antibacterial effects. In particular, doxycycline is a potent inhibitor of matrix metalloproteinase 9, which is a protease derived largely from neutrophils. Recent studies demonstrate a significant correlation between pulmonary disease severity and sputum concentrations of MMP-9 in patients with CF. In addition, sputum MMP-9 levels are associated with airway remodeling in CF.

The goal of this study is to determine the therapeutic potential of doxycycline in modulating host airway inflammation in patients with CF. Specifically, the study will characterize the PK /PD of doxycycline, evaluate the safety of short term therapy, and explore the concentration effect relationship between doxycycline exposure and sputum biomarker levels.

DETAILED DESCRIPTION:
This study will consist of a prospective, open-label, randomized, controlled trial conducted in 24 patients with cystic fibrosis. Twenty subjects will be stratified in a 1:2 ratio based on baseline FEV1 into mild (> 70%) or moderate (40-70%) pulmonary disease in order to control for disease severity within each dose level. The subjects will be randomized in blocks of four to receive no drug, 40mg, 100mg, or 200mg daily for 28 days.

Sputum samples will be obtained in all groups by induction with hypertonic saline at baseline, 8, 24, and 48 hours following the first dose and then weekly for 4 weeks. Sputum will also be collected at two follow up visits after the treatment period at weeks 5 and 6.

In the doxycycline group, serial blood samples (5 mL) for determination of doxycycline concentrations will be obtained before and at 0, 0.5, 1, 2, 4, 12, 24, and 48 hours following the 1-hr infusion of a single IV dose. Once daily dosing of doxycycline will resume immediately following the 48-hour blood sample and will continue until day 28. Additional levels will be obtained pre-dose, and 1, 2, and 3 hours after doses administered on days 14 and 28. A sample of blood will be obtained at baseline, and at days 28 for inflammatory marker analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Clinically stable (FEV1 within 10% of baseline)
* FEV1 > 40% predicted

Exclusion Criteria:

* Use of clinically significant concomitant drug therapy such as long-term use of nonsteroidal anti-inflammatory drugs or corticosteroids
* Known hypersensitivity to doxycycline
* Pregnancy or attempting to conceive, breast feeding, initiation of or change in hormonal method of contraception within 4 weeks of baseline or during the study
* Use of systemic antibiotics (except oral azithromycin) within 4 weeks of baseline
* Use of doxycycline within 60 days of baseline
* Known history of gastrointestinal bleeding or gastrointestinal ulceration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of doxycycline on inflammatory biomarkers | Within 42 days

SECONDARY OUTCOMES:
To characterize the pharmacokinetics, pharmacodynamics and safety of doxycycline in patients with cystic fibrosis | Within 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Beringer, Pharm.D., Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

REFERENCES:
- [Result] Beringer PM, Owens H, Nguyen A, Benitez D, Rao A, D'Argenio DZ. Pharmacokinetics of doxycycline in adults with cystic fibrosis. Antimicrob Agents Chemother. 2012 Jan;56(1):70-4. doi: 10.1128/AAC.05710-11. Epub 2011 Oct 24. PMID 22024822